CLINICAL TRIAL: NCT04266067
Title: The Effects of PNF and Frenkel's Exercises on Balance, Fall Risk, and Quality of Life in Postmenopausal Women
Brief Title: PNF and Frenkel's Exercises for Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Yeşil (Other)
Responsible Party: Sponsor-Investigator, Hilal Yeşil, Assoc. Prof., Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HYSS2019
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Postmenopausal Symptoms
Keywords: PNF exercise; Frenkel exercise
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF exercise (Active Comparator): In the PNF exercise group; exercises were performed in company with a physiotherapist 5 days a week (30 minutes ) for 4 weeks. Five specific techniques were applied to the patients: dynamic stabilization, rhythmic stabilization, combined isotonic contractions, and hold-relax active motion
  Interventions: Other: PNF exercise
- Frenkel exercise (Active Comparator): In the Frenkel exercise group, Frenkel coordination exercises were given in home exercise program 5 days a week for 4 weeks.The physiotherapist demonstrated Frenkel exercises to them once.
  Interventions: Other: Frenkel exercise

INTERVENTIONS:
Other: PNF exercise — Proprioceptive neuromuscular facilitation (PNF) is a form of neuromuscular retraining type containing the stimulation of sensory receptors to provide information about the body position and movement to facilitate the intended movement
  Arms: PNF exercise
Other: Frenkel exercise — The Frenkel exercises consist of a series of slow, repetitive movements performed in different positions while lying, sitting and standing.
  Arms: Frenkel exercise

SUMMARY:
Postural stability is impaired due to the decrease in estrogen in the postmenopausal period, which may lead to disruption of balance and risk of falling. Our objective was to investigate the effects of PNF and Frenkel's exercises on balance, fall risk, and quality of life in postmenopausal women.

Methods: Forty-eight postmenopausal women were randomized into PNF (n = 24) (5 days a week) and Frenkel (n = 24) (5 days a week as a home exercise program) exercise groups. Hand grip strength, quality of life (short form- 36), falling risk (Falls Risk of Older People-Community Setting [FROP-COM]), and balance (functional reach test [FRT], one - leg stand test [OLST], timed up and go test [TUG], and Berg balance scale [BBS]) of all patients were evaluated prior to treatment, and at 4th week follow-up. The treatment responses were evaluated at the beginning, and at the 4th week.

DETAILED DESCRIPTION:
In this study, we aimed to investigate the effects of PNF and Frenkel's exercises on balance, fall risk, and quality of life in postmenopausal women.

Methods: Forty-eight postmenopausal women were randomized into PNF (n = 24) (5 days a week) and Frenkel (n = 24) (5 days a week as a home exercise program) exercise groups. Hand grip strength, quality of life (short form- 36), falling risk (Falls Risk of Older People-Community Setting [FROP-COM]), and balance (functional reach test [FRT], one - leg stand test [OLST], timed up and go test [TUG], and Berg balance scale [BBS]) of all patients were evaluated prior to treatment, and at 4th week follow-up. The treatment responses were evaluated at the beginning, and at the 4th week. A total of 13 patients (27.1%) had a history of falls in the last 6 months and 12 months. According to the intra-group assessment; there was a significant improvement in all parameters in PNF group (p<0.05). In Frenkel group, there was a significant improvement in all evaluations except the OLST (p=0.064), and the short form-36 mental health score (p=0.057). Among the groups; no significant difference was detected in terms of hand grip strength, FROP-COM, FRT and TUG scores (p > 0.05). The OLST and BBS scores was significantly higher in the PNF group (p=0.022, and p= 0.002, respectively). To conclude, PNF and Frenkel exercise programs had significant effects on balance parameters, risk of falling and quality of life in postmenopausal women. Frenkel home exercise program is cheaper, easier, and requires less manpower, therefore, we think that it may be more preferable in terms of improving balance and reducing fall risk in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

- Postmenopausal women aged between 50-80 years who can walk independently were included in the study

Exclusion Criteria:

* 1. Having diabetic retinopathy and nephropathy, 2. The presence of plantar ulcers, 3. Presence of coronary artery disease, 4. Presence of peripheral vascular disease, 5. Presence of vision disorders, 6. Having a history of use of assistive walking device, 7. Presence of severe neurological, muscular or rheumatologic disease, 8. History of alcohol use, 9. Having lower limb amputation, 10. Presence of dementia, 11. Having a malignancy history, 12. Having a hearing problem, 13. Using a drug affecting balance, 14. Patients included in regular exercise program, and 15. Presence of neurological diseases affecting balance (stroke, multiple sclerosis, Parkinson's disease, epilepsy, etc.).

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Falls Risk for Older People-Community Setting (FROP-COM) score at 4 th week. | up to 4 weeks
  FROP-COM); includes 13 fall risk factor sections. The sum of the individual scores provides a total fall risk score ranging between 0 and 60 and higher scores refer to higher risks. While scores between 0-20 are evaluated as low- moderate fall risk, those between 21-60 scores are evaluated as high fall risk

SECONDARY OUTCOMES:
change from baseline Functional reach test score at 4 th week | up to 4 weeks
  Functional reach test is a performance-based test measuring the maximum distance a person can reach while standing in a fixed position without losing balance, taking a step or touching a wall. The patients were asked to reach forward as far as possible without falling and stepping. The distance between the start and end positions was measured and recorded. Three trials were conducted and the average of the last two was noted .
change from baseline one leg stand test score at 4 th week | up to 4 weeks
  One leg stand test; as the starting position, the patients were asked to stand in a relaxed way with their eyes open with evenly distributed weight on both feet. The patients were then asked to stand freely on one leg for as long as possible. The test was terminated after 30 seconds or when the patient's foot touched to the ground. Then, the time was recorded
change from baseline timed up and go test score at 4 th week | up to 4 weeks
  Timed up and go test; the patient was asked to stand up while sitting in a chair, to walk to a line three meter away at a comfortable and safe speed and then return back and sit again on the chair. In this process, time was kept with stopwatch. In order to determine fall risk, a cut-off point of ≥13.5 seconds was used
change from baseline berg balance scale score at 4 th week | up to 4 weeks
  Berg balance scale (BBS) is a scale consisting of 14 items. Each of these items is scored between 0 and 4. "0" indicates that the task cannot be done. As the score goes to 4, the patient completes the task independently. Total score range is between 0 and 56. Here, while 0 point reflect the worst balance, 56 points refer to the best balance
change from baseline hand grip strength test score at 4 th week | up to 4 weeks
  Hand grip strength test; was evaluated with JAMAR dynamometer (BASELINE hydraulic hand dynamometer FEI White Plains, NY 10602 USA). The patients were asked to sit flat, hold their upper arm in a neutral position and keep their elbows at 90° flexion. The forearm was held in a neutral position and they were asked to hold their elbow in extension between 0 and 30°. The patient was then asked to grip the device with all of his/her strength.
change from baseline short form 36 score at 4 th week | up to 4 weeks
  Short form (SF)- 36; is a generic scale frequently used to assess quality of life. SF-36 is composed of 36 items used in the calculation of 8 different scale scores and consists of the following eight subscales. While 0 point indicates the worst health status, 100 points signify best health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal Yesil, Afyonkarahisar, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No